CLINICAL TRIAL: NCT00894595
Title: Preventing Knee Injuries in Adolescent Female Football Players - Protocol of a Cluster-randomized Controlled Trial
Brief Title: Preventing Knee Injuries in Adolescent Female Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Swedish Football Association (Unknown); Folksam (Other); Swedish National Centre for Research in Sports (Unknown)
Responsible Party: Markus Waldén, MD, PhD, Linköping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M197-08
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Knee Injury
Keywords: Incidence of ACL injury; Risk factors for ACL injury; Prevention of ACL injury or any acute knee injury
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The clubs in the intervention group are instructed to perform a warm-up program at two training sessions per week throughout the entire 2009 competitive season.
  Interventions: Behavioral: Knäkontroll, SISU Idrottsböcker©, Sweden, 2005
- Control group (Active Comparator): The clubs in the control group are instructed to train and play as usual throughout the 2009 season
  Interventions: Behavioral: Knäkontroll, SISU Idrottsböcker©, Sweden, 2005

INTERVENTIONS:
Behavioral: Knäkontroll, SISU Idrottsböcker©, Sweden, 2005 — The preventive program (Knäkontroll, SISU Idrottsböcker©, Sweden, 2005) consists of six exercises focusing on knee control and core stability and is performed during the warm-up at two training sessions per week throughout the 2009 competitive season.

SUMMARY:
Football-related knee injuries are common and especially the anterior cruciate ligament (ACL) injury constitute a serious problem in football regardless of the playing level. The purpose of this study is to conduct a randomized controlled trial evaluating the effect of a training program designed to prevent acute knee injury in female adolescent football players.

The investigators' hypotheses are:

1. a preventive training program reduces the incidence of ACL injury, and
2. a high match frequency and match play at senior level increase the risk of ACL injury.

ELIGIBILITY:
Inclusion Criteria:

* Teams with female football players aged 13-17 years

Exclusion Criteria:

* Teams that did not reply to the invitation or declined participation
* Teams having less than two scheduled training sessions per week
* Teams already using the preventive program

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4564 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The incidence of ACL injury | One competitive football season

SECONDARY OUTCOMES:
The incidence of any acute knee injury except contusion | One competitive football season

CONTACTS AND LOCATIONS:
Overall Officials: Markus Waldén, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Medical and Health Sciences, Linköping University, Linköping, Sweden

REFERENCES:
- [Derived] Walden M, Atroshi I, Magnusson H, Wagner P, Hagglund M. Prevention of acute knee injuries in adolescent female football players: cluster randomised controlled trial. BMJ. 2012 May 3;344:e3042. doi: 10.1136/bmj.e3042. PMID 22556050
- [Derived] Hagglund M, Walden M, Atroshi I. Preventing knee injuries in adolescent female football players - design of a cluster randomized controlled trial [NCT00894595]. BMC Musculoskelet Disord. 2009 Jun 23;10:75. doi: 10.1186/1471-2474-10-75. PMID 19545453